CLINICAL TRIAL: NCT04723602
Title: Phase 1b Trial to Evaluate Safety, Tolerability and Immune Responses of 2 Monovalent Chimpanzee Adenoviral Vectored Filovirus (Ebola-S and Marburg) Vaccines to Healthy Adults, Collection of Plasma/Serum for the Purposes of Assay Development
Brief Title: Evaluation of Safety, Tolerability and Immune Responses of Ebola-S and Marburg Vaccines in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Albert B. Sabin Vaccine Institute (Other)
Collaborators: ICON plc (Industry); Oklahoma Blood Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Sabin 001
Record Dates: First submitted 2020-12-10; First posted 2021-01-26 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Ebola Virus Disease; Marburg Virus Disease
Keywords: Coronavirus Disease; Creatine phosphokinase; Clinical Research Associate; Contract Research Organization; Division of AIDS; Disseminated Intravascular Coagulation; Diagnostic Lab of Oklahoma; Deoxyribonucleic Acid; Species Zaire Ebolavirus; Electronic Case Report Form; Ethylenediaminetetraacetic Acid; Ebola Hemorrhagic Fever; Enzyme-Linked Immunosorbent Assay; Food and Drug Administration; Ebola Virus Disease; Degrees Fahrenheit; Good Clinical Practices; Good Laboratory Practices; Grams; Glycoprotein; Government and Public Health Solutions; GlaxoSmithKline; Hemagglutinin; Hereditary Angioedema; Hepatitis B Virus; Hepatitis C Virus; Human immunodeficiency virus; Human T-cell Leukemia Lymphoma Virus; Investigator's Brochure; International Council for Harmonisation; International Committee on the Taxonomy of Viruses; Identification; Immunoglobulin G; Immunoglobulin M; Intramuscular(ly); Investigational New Drug; Investigational product; Intravenous; Marburg Virus; Marburg Virus Disease; Marburg hemorrhagic fever; Milliliter; Millimeters of Mercury; Modified Vaccinia Ankara; Nucleic Acid Test; Non-Disclosure Agreement; Non-Human Primate; National Institute of Allergy and Infectious Diseases; National Institutes of Health; Nucleoprotein; Nonsteroidal Anti-Inflammatory Drug; Oklahoma Blood Institute; Office for Human Research Protection; Plasmapheresis Assessment Review Team; Plaque Forming Unit; Physical Exam; Principal Investigator; Post Injection Reactogenicity; Project Manager; Prothrombin Time; Partial Thromboplastin Time; Particle Units; Ravn Virus; Recombinant Human Adenovirus Serotype 5; Species Reston ebolavirus; Ribonucleic Acid; Rapid Plasma Regain; Reverse Transcription Polymerase Chain Reaction; Serious Adverse Event; Severe Acute Respiratory Syndrome Coronavirus 2; Statistical Analysis System; Schedule of Events; Standard Operating Procedure; Serum Separator Tube; Species Sudan Ebolavirus; Suspected, Unexpected and Serious Adverse Reaction; Species Taï Forest Ebolavirus; Technical Resources International, Inc; Universal Donor History Questionnaire; Upper Limit of Normal; Viral Particles; Vaccine Research Center; Vesicular Stomatitis Virus; Variant Creutzfeldt-Jakob Disease; White blood cell; World Health Organization; Western Institutional Review Board; Wild type; Zaire Ebola virus; Acquired Angioedema; Program, Inc.; Human adenovirus Serotype 5; Activities of Daily Living; Adverse Event; Acquired Immunodeficiency Syndrome; Alanine aminotransferase; Assessment of Understanding; Aspartate Aminotransferase; Biomedical Advanced Research and Development Authority; Species Bundibugyo ebolavirus; Blood Establishment Computer System; Body mass index; Blood Urea Nitrogen; Recombinant Chimpanzee Adenovirus Serotype 3; Recombinant Chimpanzee Adenovirus; Recombinant Chimpanzee Adenovirus Serotype 63; Complete blood count; Center for Disease Control and Prevention; Code of Federal Regulations; Confidence Interval; Centimeters; Type 3-Vectored Ebola virus Vaccine; Type 3-Vectored Ebola Sudan Vaccine; Type 3-Vectored Marburg Vaccine
MeSH Terms: conditions — Hemorrhagic Fever, Ebola; Marburg Virus Disease; Disseminated Intravascular Coagulation; Angioedemas, Hereditary; Hepatitis B; Hepatitis C; Acquired Immunodeficiency Syndrome; Communicable Diseases; Creutzfeldt-Jakob Syndrome; Acquired angioedema

STUDY DESIGN:
Intervention Model Description: 2 cohorts of 16 participants each.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- cAd3-Marburg at 1 x 10^11 Particle Units (PU) (Active Comparator): A total of 16 healthy adults will be enrolled and vaccinated with a single dose of vaccine. Group 1 (N = 16) will receive a single injection of cAd3-Marburg at 1 x 10^11 Particle Units (PU) vaccine.
  Interventions: Biological: cAd3-Marburg
- cAd3-EBO-S at 1 x 10^11 PU vaccine (Active Comparator): A total of 16 healthy adults will be enrolled and vaccinated with a single dose of vaccine. Group 2 (N = 16) will receive a single injection of cAd3-EBO-S at 1 x 10^11 Particle Units (PU) vaccine.
  Interventions: Biological: cAd3-EBO-S

INTERVENTIONS:
Biological: cAd3-Marburg — A total of 16 healthy adults will be enrolled and vaccinated with a single dose of vaccine. Group 1 (N = 16) will receive a single injection of cAd3-Marburg at 1 x 10^11 Particle Units (PU) vaccine.
  Arms: cAd3-Marburg at 1 x 10^11 Particle Units (PU)
Biological: cAd3-EBO-S — A total of 16 healthy adults will be enrolled and vaccinated with a single dose of vaccine. Group 2 (N = 16) will receive a single injection of cAd3-EBO-S at 1 x 10^11 Particle Units (PU) vaccine.
  Arms: cAd3-EBO-S at 1 x 10^11 PU vaccine

SUMMARY:
Primary Objective:

• To evaluate the safety and tolerability of cAd3-EBO-S and cAd3 Marburg vaccines when administered Intramuscular (IM) at a dose of 1 x 10^11 particle units (PU) to healthy adults.

Secondary Objectives:

* To evaluate the antibody response to Monovalent Chimpanzee Adenoviral Vectored Filovirus Ebola-S (cAd3-EBO-S) and Monovalent Chimpanzee Adenoviral Vectored Filovirus (Marburg) (cAd3 Marburg) vaccines as assessed by antigen glycoprotein (GP) specific (enzyme-linked immunosorbent assay) ELISA
* To collect sufficient post-vaccination plasma to support further development of filovirus assays

DETAILED DESCRIPTION:
Primary Endpoints: Safety

Assessment of product safety will include clinical observation and monitoring of clinical chemistry and hematology parameters. Safety will be closely monitored after injection and evaluated through Day 99 and one additional safety follow-up telephone call on Day 181 (± 14 Days). The following parameters will be assessed:

* Occurrence and severity of solicited local reactogenicity signs and symptoms for 7 days following the vaccination
* Occurrence and severity of solicited systemic reactogenicity signs and symptoms for 7 days following the vaccination
* Change from baseline for safety laboratory measures
* Occurrence of adverse events of all severities through 28 days after vaccination
* Occurrence of serious adverse events and new chronic medical conditions through the last safety follow up call at Day 181(± 14 days)

Secondary Endpoints :

* Antibody levels against vaccines cAd3-EBO-S and cAd3 Marburg as measured by enzyme-linked immunosorbent assay (ELISA) on Day 1, 15, 22, 29, 36, 43, 50, 57 and 64
* 20 Liters of plasma per vaccine group will be collected for the purpose of assay development

ELIGIBILITY:
Inclusion Criteria:

* Male or female participant must be between 18-50 (inclusive) years of age;
* Meet criteria for plasma donation*;
* Available for clinic follow-up through Day 99 and one additional follow-up call on Day 181 (±14 days);
* Agrees not to receive any vaccine from day of enrollment through Day 99;
* Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process;
* Agree to have photos taken of the vaccination site, if indicated ;
* Willing to complete repeated plasmapheresis and other protocol requirements;
* Must complete an Assessment of Understanding (AoU) by answering 9 out of 10 questions correctly at least once in 3 attempts;
* Willing to donate blood for sample storage and future unspecified assay development;
* Able to read (English) and willing to complete informed consent process;
* In good general health without clinically significant medical history, based on medical history, physical examination, vital signs and clinical laboratory results;
* Physical examination and laboratory results without clinically significant findings and a body mass index (BMI) ≥ 17 and ≤ 35 within the 28 days prior to vaccination;
* Laboratory Criteria within 28 days prior to vaccination (normal per testing laboratory) for: complete blood count (CBC) with differential count, alanine aminotransferase (ALT), serum creatinine and total protein;
* Serology screen negative for infectious diseases (hepatitis B, hepatitis C, HIV, HTLV (Human T-cell leukemia lymphoma virus), Chagas disease, Syphilis;
* Nucleic acid test (NAT) negative for Human Immunodeficiency Virus (HIV), Hepatitis C Virus (HCV), Hepatitis B Virus (HBV), West Nile and Zika;
* Negative antibody and reverse transcription polymerase chain reaction (RT-PCR) for severe acute respiratory syndrome Covid 2 (SARS CoV-2) and free of current or prior symptoms concerning for COVID-19. Participants with a previous positive RT-PCR, at least 90 days prior to screening as reported in medical history, will not be excluded if they are antibody negative;
* Female participant specific criteria:

  * Negative pregnancy serum test at screening and, negative urine pregnancy test before vaccination unless one of the following criteria is met:
* At least 1 year post-menopausal;
* Surgically sterile;

  * Use of oral, implantable, transdermal or injectable contraceptives for 21 days prior to and agrees to use through Day 181 ;
  * Use of another reliable form of contraception must be approved by the Investigator (e.g., double barrier method, Depo-Provera, intrauterine device, Norplant, oral contraceptives, contraceptive patches);
* Male participants must agree:

  * Not to father a child or donate sperm through Day 181;
  * To use an effective means of birth control from at least 21 days prior to enrollment through Day 181 if assessed to be of reproductive potential.

Meet the criteria described in the AABB (formerly known as American Association of Blood Bank) and Uniform Donor History Questionnaire, with the exception of travel for malaria or Variant Creutzfeldt-Jakob Disease (vCJD) risk

Exclusion Criteria:

* Investigational COVID-19, Ebola or Marburg vaccine in a prior clinical trial or prior receipt of a cAd3 adenoviral vectored investigational vaccine;

  * Use of immunomodulators and systemic glucocorticoids in daily doses of glucocorticoid equivalence > 20 mg of prednisolone in the last 90 days and for periods exceeding 10 days. Non-steroidal anti-inflammatory drugs [NSAIDS] are permitted. Participants that have used less than the stated glucocorticoid dose may still be excluded at the Investigator's discretion;
  * Blood products within 112 days prior to enrollment;
  * Investigational research agents within 90 days prior to enrollment;
  * Any licensed vaccine, inclusive of "live-attenuated" vaccine (e.g., oral polio, yellow fever, measles, etc.), killed, or subunit vaccine, within 28 days prior to enrollment;
  * Any experimental vaccines within 6 months prior to enrollment;
  * Current anti-tuberculosis prophylaxis or therapy;
* Female participant specific criteria: woman who is pregnant, breast-feeding or planning to become pregnant through Day 181 (±14 days);
* Unsatisfactory vein assessment for plasmapheresis via peripheral access (more details in Section 5.2.1)
* History of any of the following clinically significant conditions:

  * Serious adverse reactions to vaccines such as anaphylaxis, urticaria (hives), respiratory difficulty, angioedema, or abdominal pain;
  * Allergic reaction to excipients in the study vaccine including gentamycin, neomycin or streptomycin;
  * Clinically significant autoimmune disease or immunodeficiency;
  * Asthma that is not well controlled;
  * Positive result on a rapid plasma regain (RPR) test (A blood test for Syphilis);
  * Diabetes mellitus Type I or II;
  * Thyroid disease that is not well controlled ;
  * A history of hereditary angioedema (HAE), acquired angioedema (AAE), or idiopathic forms of angioedema;
  * Idiopathic urticaria within the last 1 year;
  * Hypertension that is not well controlled;
  * Bleeding disorder diagnosed by a doctor or use of anticoagulant medications such as, Coumadin, Eliquis, Pradaxa (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws;
  * A malignancy that is active, currently being treated, or not surgically cured (breast or prostate cancer successfully treated, with or without surgery is excluded; if diagnosed malignancy is 5 or more years prior to enrollment and cured with no ongoing treatment it will NOT be considered an exclusion);
  * Seizure in the past 3 years or treatment for seizure disorder in the past 3 years;
  * Asplenia or functional asplenia;
  * Psychiatric condition that precludes compliance with the protocol; past or present psychoses; or within five years prior to enrollment, history of a suicide plan or attempt;
  * Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a participant's ability to give informed consent.
  * Abnormal laboratory results (per testing laboratory)
  * Positive COVID-19 symptom screen, SARS-CoV-2 RT-PCR, or SARS CoV-2 antibody test

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
Safety of Ebola and Marburg vaccines assessed by clinical observation. | 7 Days
  Safety of Ebola and Marburg vaccines, as seen in local reactogenicity signs and symptoms with diary questionnaire card.
Safety of Ebola and Marburg vaccines assessed by clinical observation. | 7 Days
  Safety of Ebola and Marburg vaccines, as seen in systemic reactogenicity signs and symptoms with diary questionnaire card.
Safety of Ebola and Marburg vaccines assessed by change from baseline in levels of Complete Blood Count (CBC). | 6 months
  Safety of Ebola and Marburg vaccines assessed by change in levels of Complete Blood Count (CBC) w/differential count as laboratory measures of safety from baseline.
Safety of Ebola and Marburg vaccines assessed by change from baseline in levels of Creatinine. | 6 months
  Safety of Ebola and Marburg vaccines assessed by change in levels of Creatinine as laboratory measures of safety from baseline.
Safety of Ebola and Marburg vaccines assessed by change from baseline in levels of Alanine Transaminase (ALT). | 6 months
  Safety of Ebola and Marburg vaccines assessed by change in levels of Alanine Transaminase (ALT) as laboratory measures of safety from baseline.
Safety of Ebola and Marburg vaccines assessed by adverse experiences. | 28 days
  Safety of Ebola and Marburg vaccines assessed by adverse events of all severities (Mild, moderate, and severe)
Safety of Ebola and Marburg vaccines assessed by serious adverse experiences. | 6 months
  Safety of Ebola and Marburg vaccines assessed by serious adverse events of all severities (Mild, moderate, and severe)

SECONDARY OUTCOMES:
Evaluation of antibody response to cAd3-EBO-S and cAd3 Marburg vaccines | Measured at Day 1, 15, 22, 29, 36, 43, 50, 57, and 64
  Immunogenicity of the Ebola and Marburg vaccines as measured by antigen GP-specific ELISA
Collection of sufficient post-vaccination plasma to support further development of filovirus assays. | May be collected at Day 29, 36, 43, 50, 57 and/or 64
  20 L of plasma per vaccine group (N=2) will be collected for the purpose of assay development. 800 mL of plasma will be collected at Day 29. Thereafter, plasma collections will be up to approximately 600 mL. Participants may donate up to 6 total times and all collections will be done within the limits of the FDA approved instructions for use for the Fenwal Alyx collection device.

CONTACTS AND LOCATIONS:
Overall Officials: Roxana Rustomjee, MBChB, Study Chair — The Albert B. Sabin Vaccine Institute; Michael Stevenson, MD, Principal Investigator — Oklahoma Blood Institute; David Hoover, MD, Study Director — ICON plc; Tuan Le, MD, Principal Investigator — Oklahoma Blood Institute
Locations (1):
- Oklahoma Blood Institute (OBI), Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sanchez A, Kiley MP, Klenk HD, Feldmann H. Sequence analysis of the Marburg virus nucleoprotein gene: comparison to Ebola virus and other non-segmented negative-strand RNA viruses. J Gen Virol. 1992 Feb;73 ( Pt 2):347-57. doi: 10.1099/0022-1317-73-2-347. PMID 1538192
- [Result] Sanchez A, Kiley MP, Holloway BP, Auperin DD. Sequence analysis of the Ebola virus genome: organization, genetic elements, and comparison with the genome of Marburg virus. Virus Res. 1993 Sep;29(3):215-40. doi: 10.1016/0168-1702(93)90063-s. PMID 8237108
- [Result] Geisbert TW, Jahrling PB. Exotic emerging viral diseases: progress and challenges. Nat Med. 2004 Dec;10(12 Suppl):S110-21. doi: 10.1038/nm1142. PMID 15577929
- [Result] Hensley LE, Jones SM, Feldmann H, Jahrling PB, Geisbert TW. Ebola and Marburg viruses: pathogenesis and development of countermeasures. Curr Mol Med. 2005 Dec;5(8):761-72. doi: 10.2174/156652405774962344. PMID 16375711
- [Result] Ledgerwood JE, DeZure AD, Stanley DA, Coates EE, Novik L, Enama ME, Berkowitz NM, Hu Z, Joshi G, Ploquin A, Sitar S, Gordon IJ, Plummer SA, Holman LA, Hendel CS, Yamshchikov G, Roman F, Nicosia A, Colloca S, Cortese R, Bailer RT, Schwartz RM, Roederer M, Mascola JR, Koup RA, Sullivan NJ, Graham BS; VRC 207 Study Team. Chimpanzee Adenovirus Vector Ebola Vaccine. N Engl J Med. 2017 Mar 9;376(10):928-938. doi: 10.1056/NEJMoa1410863. Epub 2014 Nov 26. PMID 25426834